CLINICAL TRIAL: NCT00121147
Title: A Comparison of the Additivity of Brinzolamide Ophthalmic Suspension, 1% (Azopt) and Brimonidine Tartrate Ophthalmic Solution, 0.15% (Alphagan P) to Travoprost Ophthalmic Solution, 0.004% (Travatan) in Patients With Elevated IOP on Travoprost. A Three Month Double-Masked, Multi-Center Trial in the United States
Brief Title: Additivity Study: Additive Effect on Eye Pressure of Azopt and Alphagan P to Travatan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hermann Eye Center (Other)
Collaborators: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEF-042
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2006-02-24 (Estimated); Status verified 2005-07

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension; Pseudoexfoliation Syndrome
Keywords: glaucoma; pseudoexfoliation
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Exfoliation Syndrome; Glaucoma | interventions — Travoprost; brinzolamide; Brimonidine Tartrate

INTERVENTIONS:
Drug: Travatan
Drug: Azopt
Drug: Alphagan P

SUMMARY:
The purpose of this study is to compare the additive effect on eye pressure of Azopt and Alphagan P to Travatan.

DETAILED DESCRIPTION:
The purpose of this research study is to compare the effect on the pressure inside the eye when Brinzolamide Ophthalmic Suspension, 1% (Azopt), a carbonic anhydrase inhibitor, and Brimonidine Tartrate Ophthalmic Solution, 0.15% (Alphagan-P), an alpha 2 agonist, are added to Travoprost Ophthalmic Solution, 0.004% (Travatan), a prostaglandin, in patients with primary open angle glaucoma, ocular hypertension and pseudoexfoliation syndrome. Brinzolamide Ophthalmic Suspension, 1% (Azopt), Brimonidine Tartrate Ophthalmic Solution, 0.15% (Alphagan-P), and Travoprost Ophthalmic Solution, 0.004% (Travatan) are all currently approved by the FDA and on the market, being used by patients. Even though all three medications are currently approved for the purpose of the study they will be considered study medicines.

Glaucoma, Ocular Hypertension and Pseudoexfoliation syndrome have been treated with IOP-lowering medications or surgery to lower the pressure inside the eye to reduce the risk of visual field loss. Today, common treatments for a patient often begins with the prescription of a prostaglandin (Travoprost). If the prostaglandin does not lower the pressure inside the eye enough, a second drug is usually added. Topical carbonic anhydrase inhibitors (Brinzolamide) and alpha 2 agonists (Brimonidine) are common choices as additive medicines.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age: 35 years
* Uni or bilateral primary open angle glaucoma, ocular hypertension or pseudoexfoliation syndrome (POAG is defined as having VF and optic nerve changes consistent with glaucomatous disease)
* Insufficient response to monotherapy: defined as IOP > 18mm Hg (mean diurnal) and less than 32 mm Hg on Travatan at baseline
* Informed consent and HIPPA consent obtained at screening visit prior to any study events
* Ability to adhere to study treatment visit plan

Exclusion Criteria:

* Closed, occluded, or potentially occludable angle
* History of angle closure
* Previous intraocular surgery, except uncomplicated clear cornea phacoemulsification or argon laser trabeculoplasty
* Argon laser trabeculoplasty or phacoemulsification within the last 3 months
* Central corneal thickness outside the 500 - 600 (inclusive) micron range as measured by ultrasonic pachymetry
* Ocular or periocular inflammation within 3 months prior to study (except blepharitis related or seasonal allergic conjunctivitis)
* History of uveitis or previous intraocular inflammation (other than post-operatively)
* Hypersensitivity to sulfa, alpha agonists or benzalkonium chloride
* History of use of any steroids for over 1 week within 3 months of screening or likely need for any corticosteroids during the study (except inhaled, nasal or topical non-ocular)
* Use of systemic medications known to effect IOP (e.g. Alpha agonists, Beta blockers, Ace inhibitors and angiotensin II receptor blockers) which have not been stable for three months prior to baseline and the dosage is not expected to change during the course of the study

Women

* Pregnancy (study medications have been determined to cause possible harm to the fetus)
* Women of childbearing potential who are not using contraceptive methods. Childbearing potential is defined as any woman who is not postmenopausal (12 months without a menstrual period) or surgically sterile. Contraceptive methods are defined as abstinence, having a vasectomized partner, or ongoing use of approved oral, injectable, topical or implanted contraceptives, a barrier method or an IUD

General:

* Use of any investigational medication within one month prior to baseline visit

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-09; Study Completion 2005-10

PRIMARY OUTCOMES:
Mean decrease in diurnal intraocular pressure (IOP) (mean of the three daily intraocular pressures) at month 3 visit

SECONDARY OUTCOMES:
Change in IOP from baseline at each time point
IOP at 8AM (prior to dosing), 12 noon and 4 pm at month 3
Percent IOP lowering from pretreatment baseline to the three month visit. Both diurnal average and at each time point
Percent of patients reaching specific target pressures after three months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Feldman, M.D., Study Chair — Hermann Eye Fund / University of Texas
Locations (21):
- United States (21):
  - Doheny Eye Institute, Los Angeles, California
  - The Eye Center, Hamden, Connecticut
  - University of Florida, Gainesville, Florida
  - Emory Healthcare Eye Center, Atlanta, Georgia
  - Omni Eye Services, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois Eye and Ear Infirmary, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Glaucoma Consultation Service, Boston, Massachusetts
  - Kresge Eye Institute, Detroit, Michigan
  - Mississippi Eye Associates, Ocean Springs, Mississippi
  - Eyecare Ophthalmology PC, Bethpage, New York
  - Mount Sinai School of Medicine, New York, New York
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Wills Eye Institute, Philadelphia, Pennsylvania
  - The Keystone Eye Associates, Philadelphia, Pennsylvania
  - Glaucoma Associates of Texas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Hermann Eye Center, Houston, Texas
  - Lone Star Eye Associates, Sugarland, Texas
  - West Virginia University Eye Institute, Morgantown, West Virginia